CLINICAL TRIAL: NCT03701802
Title: Immunogenetic Modulators of Mucosal Protection From HIV-1: The Kinga Study
Brief Title: Immunogenetic Modulators of Mucosal Protection From HIV-1
Acronym: Kinga
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Kenya Medical Research Institute (Other)
Responsible Party: Principal Investigator, Jairam Lingappa, Professor, University of Washington
Other Study IDs: STUDY00001559; R01AI129715 (NIH); R01AI131914 (NIH); R01AI141435 (NIH)
Record Dates: First submitted 2018-09-21; First posted 2018-10-10 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: HIV Infections; HSV-2 Infection
Keywords: HIV prevention; Tenofovir Disoproxil Fumarate (TDF)/Emtricitabine (FTC); PrEP
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Genital samples Blood samples Urine samples Saliva samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HIV-1 serodiscordant couples: Heterosexual couples in which one partner is infected with HIV-1 and the other partner is HIV-1 uninfected
- Concordant HIV-1 negative couples: Heterosexual couples in which both partners are HIV-1 uninfected

SUMMARY:
This is a single site, prospective, observational study that seeks to assess changes in mucosal immunity that occur as a result of HIV-1 exposure, HSV-2 infection, and/or pre-exposure prophylaxis (PrEP) usage to prevent HIV-1 acquisition. The study will collect mucosal and peripheral blood samples for a detailed analysis of longitudinal immune responses, while also obtaining samples for genetic characterization to understand how variants in CD101 and UBE2V1 may modulate host mucosal responses and HIV-1 infection risk.

DETAILED DESCRIPTION:
A challenge to development of HIV-1 vaccines is to better understand the natural immune mechanisms for protection from HIV-1 infection. To this end, immunologists have increasingly appreciated the importance of regulatory T cells in peripheral blood that modulate the magnitude and characteristics of the host inflammatory response including against infectious diseases. The investigators have recently identified specific host genetic variants in the genes CD101 and UBE2V1 that appear to strongly predispose to HIV-1 infection risk and may act through regulatory T cells and other immunologic pathways. Most studies of individuals who are repeatedly HIV-1 exposed but remain seronegative (HESN) have focused on immunological correlates in peripheral blood rather than mucosal immune responses. However, with genital mucosal tissues being the portal of entry for heterosexually transmitted HIV-1 infection, it is critical to understand the role of immunological responses to HIV-1 that occur in the genital mucosa. A valuable model to carry out such studies is offered by evaluation of HIV-Exposed SeroNegative (HESN) individuals, particularly in the context of heterosexual sex with a stable HIV-1 infected partner e.g., HIV-1 serodiscordant couples (SDC). In order to understand how genital exposure to HIV-1 may modulate these immune pathways, HIV-1 serodiscordant couples should be compared to heterosexual partners in concordant HIV-1 negative couples (CNC) where neither partner has HIV-1. This study seeks to address this important knowledge gap by enrolling high-risk HESN with defined heterosexual HIV-1 exposures in the context of serodiscordant partnerships compared to unexposed concordant seronegative controls. The study will prospectively collect mucosal and peripheral blood samples for a detailed analysis of longitudinal immune responses, while also obtaining samples for genetic characterization to understand how variants in CD101 and UBE2V1 may modulate host mucosal responses and HIV-1 infection risk.

Primary Objectives:

* To identify mucosal immunoregulatory mechanisms mediating host response to heterosexual exposure to HIV-1.
* To determine how high priority variants in CD101 and UBE2V1 modify host mucosal responses in HIV-1 exposure and infection.

Secondary Objectives:

* Identify factors (including HIV-1 exposure, host genetic and microbiota) that modify immunoregulatory mechanisms mediating host response to HIV-1
* Evaluate how these immunogenetic regulatory mechanisms influence other infectious and immunological outcomes
* Evaluate the effect of PrEP on early HIV-1 disease

ELIGIBILITY:
Inclusion criteria:

HIV-1 Uninfected Participants;

* Age ≥18 and ≤65 and able to provide independent informed consent for research per local regulations and guidelines
* Able and willing to provide written informed consent to be screened for and to take part in the study
* Part of a heterosexual couple in which either one or both partners meet the study eligibility criteria for partner (HIV-1 uninfected) participants. Couples are defined by the following criteria:
* Partners are sexually active (defined as having had vaginal intercourse with the enrolled partner at least 6 times in the last three months)
* Partners plan to remain in the relationship for the duration of the study period.
* HIV-1 uninfected status is based on parallel negative HIV-1 rapid tests, both at study screening and at the enrollment visit
* Able and willing to provide adequate locator information for study retention purposes, as defined by local standard operating procedures

HIV-1 Infected Participants;

* Of legal age to provide independent informed consent for research per local regulations and guidelines.
* Able and willing to provide written informed consent to be screened for and to take part in the study.
* Part of a heterosexual couple in which one partner meets the study eligibility criteria for index (HIV-1 infected) participants and the other partner meets the study eligibility criteria for partner (HIV-1 uninfected) participants
* Current or previous use of antiretroviral therapy with unsuppressed HIV-1 viral load
* HIV-1 infected based on positive EIA and, when available, detectable viral load.
* No history of any clinical AIDS-defining diagnoses.
* Able and willing to provide adequate locator information for study retention purposes, as defined by local standard operating procedures.

Exclusion criteria:

HIV-1 Uninfected Participants;

* Abnormal serum creatinine (based on sub-Saharan African normal values)
* Active and serious infections, including active tuberculosis infection or osteomyelitis and all infections requiring parenteral antibiotic therapy; active clinically significant medical problems including cardiac disease, pulmonary disease, diabetes requiring hypoglycemic medication; and previously diagnosed malignancy expected to require further treatment.
* Receiving ongoing therapy with any of the following at the time of enrollment: antiretroviral therapy (ART), including nucleoside analogs, nonnucleoside reverse transcriptase inhibitors, protease inhibitors or investigational antiretroviral agents, interferon (alpha, beta, or gamma) or interleukin (e.g., IL-2) therapy, metformin, aminoglycoside antibiotics, amphotericin B, cidofovir, systemic chemotherapeutic agents, other agents with significant nephrotoxic potential, other agents that may inhibit or compete for elimination via active renal tubular secretion (e.g., probenecid), and/or other investigational agent
* At enrollment, has any other condition that, based on the opinion of the investigator or designee, would preclude provision of informed consent; make participation in the study unsafe; complicate interpretation of study outcome data)
* Pregnant at the time of screening

HIV-1 Infected Participants;

* Current or previous use of antiretroviral therapy with suppressed HIV-1 viral load
* Currently enrolled in another HIV-1 treatment trial
* At enrollment, has any other condition that, based on the opinion of the investigator or designee, would preclude provision of informed consent; make participation in the study unsafe; complicate interpretation of study outcome data; or otherwise interfere with achieving the study objectives.
* Pregnant at the time of screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: African heterosexual HIV-serodiscordant (SDC) and HIV-1 concordant negative couples (CNC)
Sampling Method: Non-Probability Sample
Enrollment: 812 (Actual)
Dates: Start 2018-09-27 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of genital-tract tissue resident memory (TRM) cells | At 6 months of follow-up
  We will compare frequency of CD69+ among CD8+ TRM in genital tissues between HIV-1 exposed and HIV-1 unexposed individuals

SECONDARY OUTCOMES:
Prevalence of genital-tract tissue resident memory (TRM) cells in individuals with versus without CD101 immunoglobulin-like (Ig-like) variants. | At 6 months of follow-up
  We will compare frequency of CD69+ among CD8+ TRM in genital tissues in individuals with versus without CD101 immunoglobulin-like (Ig-like) variants.

OTHER OUTCOMES:
Prevalence of genital-tract tissue resident memory (TRM) cells | At enrollment
  We will compare frequency of CD69+ among CD8+ TRM in genital tissues between HIV-1 exposed and HIV-1 unexposed individuals
Prevalence of genital-tract tissue resident memory (TRM) cells in individuals with versus without CD101 immunoglobulin-like (Ig-like) variants. | At enrollment
  We will compare frequency of CD69+ among CD8+ TRM in genital tissues in individuals with versus without CD101 immunoglobulin-like (Ig-like) variants.

CONTACTS AND LOCATIONS:
Overall Officials: Jairam Lingappa, MD, PhD, Study Chair — University of Washington
Locations (1):
- Partners in Health, Research and Development, Thika, Kenya

IPD SHARING:
Plan to Share IPD: Undecided
De-identified individual participant data for all outcome measures

REFERENCES:
- [Background] Pattacini L, Baeten JM, Thomas KK, Fluharty TR, Murnane PM, Donnell D, Bukusi E, Ronald A, Mugo N, Lingappa JR, Celum C, McElrath MJ, Lund JM; Partners PrEP Study Team. Regulatory T-Cell Activity But Not Conventional HIV-Specific T-Cell Responses Are Associated With Protection From HIV-1 Infection. J Acquir Immune Defic Syndr. 2016 Jun 1;72(2):119-28. doi: 10.1097/QAI.0000000000000919. PMID 26656786
- [Background] Pattacini L, Murnane PM, Baeten JM, Fluharty TR, Thomas KK, Bukusi E, Katabira E, Mugo N, Donnell D, Lingappa JR, Celum C, Marzinke M, McElrath MJ, Lund JM; Partners PrEP Study Team. Antiretroviral Pre-Exposure Prophylaxis Does Not Enhance Immune Responses to HIV in Exposed but Uninfected Persons. J Infect Dis. 2015 Jun 15;211(12):1943-52. doi: 10.1093/infdis/jiu815. Epub 2014 Dec 17. PMID 25520426
- [Background] Lund JM, Broliden K, Pyra MN, Thomas KK, Donnell D, Irungu E, Muwonge TR, Mugo N, Manohar M, Jansson M, Mackelprang R, Marzinke MA, Baeten JM, Lingappa JR. HIV-1-Neutralizing IgA Detected in Genital Secretions of Highly HIV-1-Exposed Seronegative Women on Oral Preexposure Prophylaxis. J Virol. 2016 Oct 14;90(21):9855-9861. doi: 10.1128/JVI.01482-16. Print 2016 Nov 1. PMID 27558421
- [Background] Alimonti JB, Koesters SA, Kimani J, Matu L, Wachihi C, Plummer FA, Fowke KR. CD4+ T cell responses in HIV-exposed seronegative women are qualitatively distinct from those in HIV-infected women. J Infect Dis. 2005 Jan 1;191(1):20-4. doi: 10.1086/425998. Epub 2004 Dec 1. PMID 15592998
- [Background] Biasin M, Piacentini L, Lo Caputo S, Naddeo V, Pierotti P, Borelli M, Trabattoni D, Mazzotta F, Shearer GM, Clerici M. TLR activation pathways in HIV-1-exposed seronegative individuals. J Immunol. 2010 Mar 1;184(5):2710-7. doi: 10.4049/jimmunol.0902463. Epub 2010 Feb 1. PMID 20124101
- [Background] Pattacini L, Murnane PM, Kahle EM, Bolton MJ, Delrow JJ, Lingappa JR, Katabira E, Donnell D, McElrath MJ, Baeten JM, Lund JM. Differential regulatory T cell activity in HIV type 1-exposed seronegative individuals. AIDS Res Hum Retroviruses. 2013 Oct;29(10):1321-9. doi: 10.1089/AID.2013.0075. Epub 2013 Jul 30. PMID 23815575
- [Background] Mackelprang RD, Baeten JM, Donnell D, Celum C, Farquhar C, de Bruyn G, Essex M, McElrath MJ, Nakku-Joloba E, Lingappa JR; Partners in Prevention HSV/HIV Transmission Study Team. Quantifying ongoing HIV-1 exposure in HIV-1-serodiscordant couples to identify individuals with potential host resistance to HIV-1. J Infect Dis. 2012 Oct;206(8):1299-308. doi: 10.1093/infdis/jis480. Epub 2012 Aug 27. PMID 22926009
- [Background] Wald A, Link K. Risk of human immunodeficiency virus infection in herpes simplex virus type 2-seropositive persons: a meta-analysis. J Infect Dis. 2002 Jan 1;185(1):45-52. doi: 10.1086/338231. Epub 2001 Dec 14. PMID 11756980
- [Background] Eichhorn EJ, Tandon PK, DiBianco R, Timmis GC, Fenster PE, Shannon J, Packer M. Clinical and prognostic significance of serum magnesium concentration in patients with severe chronic congestive heart failure: the PROMISE Study. J Am Coll Cardiol. 1993 Mar 1;21(3):634-40. doi: 10.1016/0735-1097(93)90095-i. PMID 8436744
- [Background] Mackelprang RD, Bamshad MJ, Chong JX, Hou X, Buckingham KJ, Shively K, deBruyn G, Mugo NR, Mullins JI, McElrath MJ, Baeten JM, Celum C, Emond MJ, Lingappa JR; Partners in Prevention HSV/HIV Transmission Study and the Partners PrEP Study Teams. Whole genome sequencing of extreme phenotypes identifies variants in CD101 and UBE2V1 associated with increased risk of sexually acquired HIV-1. PLoS Pathog. 2017 Nov 6;13(11):e1006703. doi: 10.1371/journal.ppat.1006703. eCollection 2017 Nov. PMID 29108000
- [Background] Hughes JP, Baeten JM, Lingappa JR, Magaret AS, Wald A, de Bruyn G, Kiarie J, Inambao M, Kilembe W, Farquhar C, Celum C; Partners in Prevention HSV/HIV Transmission Study Team. Determinants of per-coital-act HIV-1 infectivity among African HIV-1-serodiscordant couples. J Infect Dis. 2012 Feb 1;205(3):358-65. doi: 10.1093/infdis/jir747. Epub 2012 Jan 11. PMID 22241800
- [Background] Baeten JM, Donnell D, Ndase P, Mugo NR, Campbell JD, Wangisi J, Tappero JW, Bukusi EA, Cohen CR, Katabira E, Ronald A, Tumwesigye E, Were E, Fife KH, Kiarie J, Farquhar C, John-Stewart G, Kakia A, Odoyo J, Mucunguzi A, Nakku-Joloba E, Twesigye R, Ngure K, Apaka C, Tamooh H, Gabona F, Mujugira A, Panteleeff D, Thomas KK, Kidoguchi L, Krows M, Revall J, Morrison S, Haugen H, Emmanuel-Ogier M, Ondrejcek L, Coombs RW, Frenkel L, Hendrix C, Bumpus NN, Bangsberg D, Haberer JE, Stevens WS, Lingappa JR, Celum C; Partners PrEP Study Team. Antiretroviral prophylaxis for HIV prevention in heterosexual men and women. N Engl J Med. 2012 Aug 2;367(5):399-410. doi: 10.1056/NEJMoa1108524. Epub 2012 Jul 11. PMID 22784037
- [Derived] MacLean F, Tsegaye AT, Graham JB, Swarts JL, Vick SC, Potchen NB, Cruz Talavera I, Warrier L, Dubrulle J, Schroeder LK, Saito A, Mar C, Thomas KK, Mack M, Sabo MC, Chohan BH, Ngure K, Mugo NR, Lingappa JR, Lund JM; Kinga Study Team. Bacterial vaginosis associates with dysfunctional T cells and altered soluble immune factors in the cervicovaginal tract. J Clin Invest. 2025 Mar 25;135(10):e184609. doi: 10.1172/JCI184609. eCollection 2025 May 15. PMID 40131862
- See also: Mackelprang et. al. ftPiPHHTaPP. Rare host genetic variation influencing risk of heterosexual HIV-1 acquisition. Congress on Retroviruses and Opportunistic Infections (CROI - 2016) — http://www.croiwebcasts.org/console/player/29485?mediaType=audio&